CLINICAL TRIAL: NCT03537950
Title: Shifting Brain Excitation-Inhibition Balance Through the Endocannabinoid System in Men With Autism Spectrum Disorder (ASD) and in Healthy Controls
Brief Title: Shifting Brain Excitation-Inhibition Balance in Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Grainne McAlonan, Deputy head of department, King's College London
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HR15-162744
Record Dates: First submitted 2018-04-17; First posted 2018-05-25 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Cannabidiol; Cannabidivarin; E-I balance; pharmacological imaging
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Cannabidiol; cannabidivarin

STUDY DESIGN:
Intervention Model Description: Repeated-measures cross-over study, where each subject received each of three pharmacological probes once (order of drug administration was pseudorandomised)
Who Masked: Participant, Investigator
Masking Description: Participants and investigators were blinded to the drug condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- PLC, CBD, CBDV (Experimental): Dose order: PLC, CBD, CBDV
  Interventions: Drug: PLC; Drug: CBD; Drug: CBDV
- PLC, CBDV, CBD (Experimental): Dose order: PL, CBDV, CBD
  Interventions: Drug: PLC; Drug: CBD; Drug: CBDV
- CBD, PLC, CBDV (Experimental): Dose order: CBD, PLC, CBDV
  Interventions: Drug: PLC; Drug: CBD; Drug: CBDV
- CBD, CBDV, PLC (Experimental): Dose order: CBD, CBDV, PLC
  Interventions: Drug: PLC; Drug: CBD; Drug: CBDV
- CBDV, PLC, CBD (Experimental): Dose order: CBDV, PLC, CBD
  Interventions: Drug: PLC; Drug: CBD; Drug: CBDV
- CBDV, CBD, PLC (Experimental): Dose order: CBDV, CBD, PLC
  Interventions: Drug: PLC; Drug: CBD; Drug: CBDV

INTERVENTIONS:
Drug: PLC — Single oral dose of PLC.
  Other Names: Placebo
Drug: CBD — Single oral dose of cannabidiol (CBD) - 600mg.
  Other Names: Cannabidiol
Drug: CBDV — Single oral dose of cannabidivarin (CBDV) - 600mg.
  Other Names: Cannabidivarin

SUMMARY:
This study investigates brain response to single acute dose of cannabidiol, cannabidivarin, and placebo in healthy men with and without autism spectrum disorder

DETAILED DESCRIPTION:
Previous research suggests that cannabidiol (CBD) and cannabidivarin (CBDV) could have the potential to shift brain excitation and inhibition (E-I) in the healthy brain and in neurodevelopmental psychiatric conditions, where this balance is disrupted, such as autism spectrum disorder (ASD). However, no study to date has investigated this. Therefore, in this study, we invited 20 healthy men with and without ASD. Each participant received each drug once (600mg CBD/CBDV, or matched placebo) and magnetic resonance imaging was used to obtain measures of brain biochemistry, activity, and connectivity. We further obtained questionnaires, task data, saliva, urine and blood samples, and conducted visual tasks using eye tracking, electroencephalography, and retinal imaging.

ELIGIBILITY:
Inclusion Criteria:

* men
* pass diagnostic threshold for ASD on the ADI-R (if informant is available)
* currently symptomatic on ADOS
* age 18-50 years
* can give informed consent
* IQ>70 (on a standard instrument such as WASI)
* medication-free in the month preceding participation (but regular medication with drug, which does not affect glutamate or GABA directly may be permitted)
* willing to provide urine samples to screen for use of illicit substances prior to each scan

Exclusion Criteria:

* IQ<70
* history of psychosis, co-morbid major mental illness, significant physical illness (heart disease, high blood pressure, seizures)
* habitual substance misuse (including alcohol)
* known allergy to cannabis
* ASD caused by a known genetic syndrome e.g. Fragile X or 22q11 deletion syndrome,
* past/present treatment for epilepsy
* Women will be excluded from this pilot study to reduce heterogeneity in a small sample; avoid the issues around exposing women of reproductive age to a drug; and because pregnancy is a routine exclusion criteria for research MRI. Lastly, ASD is more common in men.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2017-02-16 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Brain biochemistry response to pharmacological stimulation | In the months 1-2 following the last day of scanning.
  The measure of brain biochemistry response to PLC, CBD, and CBDV includes the following:
  Assessment of the ratio of brain excitation and inhibition (measured as the balance of excitatory and inhibitory neurotransmitters) using using proton magnetic resonance spectroscopy [1H]MRS.

SECONDARY OUTCOMES:
Measurement of low frequency brain activity using resting state fMRI | In the months 3-4 following the last day of scanning
  In the third and fourth month following the day of the last scan, we will measure whole brain low frequency brain activity using resting state functional magnetic resonance imaging. Measure of activity: fractional amplitude of low frequency fluctuations.
Measurement of brain functional connectivity using resting state fMRI | In the months 5-6 following the last day of scanning
  In the fifth and sixth month following the day of the last scan, we will measure whole brain resting state functional connectivity using resting state functional magnetic resonance imaging. Measure of connectivity: correlation between pairs of regions.

CONTACTS AND LOCATIONS:
Overall Officials: Grainne McAlonan, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pretzsch CM, Floris DL, Voinescu B, Elsahib M, Mendez MA, Wichers R, Ajram L, Ivin G, Heasman M, Pretzsch E, Williams S, Murphy DGM, Daly E, McAlonan GM. Modulation of striatal functional connectivity differences in adults with and without autism spectrum disorder in a single-dose randomized trial of cannabidivarin. Mol Autism. 2021 Jul 1;12(1):49. doi: 10.1186/s13229-021-00454-6. PMID 34210360